CLINICAL TRIAL: NCT02575274
Title: Regenerative Treatment of Peri-Implantitis: Double Blind Randomized Controlled Clinical Trial
Brief Title: Peri-Implantitis Surgical Treatment an RCT Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mr. Sergio Diniz Ferreira (Other)
Responsible Party: Sponsor-Investigator, Mr. Sergio Diniz Ferreira, PhD student, Federal University of Minas Gerais
Organization: Federal University of Minas Gerais (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT peri-implantitis
Record Dates: First submitted 2015-01-29; First posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Peri-implantitis
Keywords: Peri-implantitis; Peri-implant disease; Dental implants; Guided bone regeneration
MeSH Terms: conditions — Peri-Implantitis | interventions — Surgical Flaps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JHS COL-HAP91 + JHS HAP-91 (Experimental): Surgical flaps debridement with plastic curette Implacare Hu-Friedy, cleaning the surface with chlorhexidine gel 2% 3 minutes and irrigation with saline solution 0.9 %. Bone defects will be treated with JHS COL-HAP91 (porous hydroxyapatite + collagen) + JHS HAP-91 (porous hydroxyapatite). Amoxicillin 500 mg 3 times/day 7 days, Tylenol 750 mg 3 times/day, and Nimesulide 100 mg 2 times/day will be prescribed.
  Interventions: Procedure: Surgical flaps
- surgical and mechanical debridement (Other): Surgical flaps: All groups will receive the same surgical treatment for implant surface decontamination. Surgical intervention will be performed with full thickness mucoperiosteal flaps. Debridement with plastic curette Implacare Hu-Friedy, cleaning the surface with chlorhexidine gel 2% 3 minutes and irrigation with saline solution 0.9 %. Amoxicillin 500 mg 3 times/day 7 days, Tylenol 750 mg 3 times/day and Nimesulide 100 mg 2 times/day will be prescribed.
  Interventions: Procedure: Surgical flaps

INTERVENTIONS:
Procedure: Surgical flaps — Surgical intervention will be performed with full thickness mucoperiostal flaps to obtain access in the bone defects. All groups will receive the same treatment for implant surface decontamination: debridement with plastic curette Implacare Hu-Friedy®, cleaning the surface with chlorhexidine gel 2% during 3 minutes and abundant irrigation with saline solution 0.9%.

SUMMARY:
The purpose of this experimental study in humans is to evaluate and compare, the regenerative therapy for the treatment of peri-implantitis using different bone substitutes and absorbable membranes with surgical therapy without the use of materials for regeneration.

DETAILED DESCRIPTION:
Specifics aims

* Compare radiographic and clinical results of guided bone regeneration (GBR) technique in the treatment of peri-implantitis using membrane and bone substitute (JHS HAP91 ® + JHS COL-HAP-91®) to surgical approach without bone substitutes.
* Compare the radiographic and clinical results of GBR with surgical therapy without biomaterials
* Evaluate radiographic changes in bone levels after GBR therapy.
* Evaluate changes in probing depth (PD) after GBR therapy.
* Evaluate the long term predictability of GBR and surgical therapy in the treatment of peri-implantitis.

Study Design This prospective clinical trial will recruit to clinical periodontal and peri-implant examination, individuals diagnosed with peri-implantitis who fit the eligibility criteria described below. After the clinical examination the individuals will receive oral hygiene instructions and those diagnosed with peri-implantitis will take implants standardized radiographic exams prior to surgery. Only circular and/or bowl-shaped bone defects will be selected for the study.

Sampling In this design the inclusion of at least 15 individuals is estimated for each experimental group when it performs a sample calculation with power of 90% and a significance level of 95% considering an outcome data from previous studies.

Individuals diagnosed with peri-implantitis will be recruited in two specialized private treatment centers and post graduation schools from June 2013 to June 2016. The total sample of 15 eligible implants with peri-implantitis per group will be treated (n total = 30).

Randomization process After the clinical and radiographic examination individuals will be scheduled for completion of the surgical procedure. It will be carried out a process of "Central Stratified Randomization" which shall consist of forty five opaque envelopes, where it will be placed the IDs of each treatment group (group 1 or group 2). The envelopes shall be sealed and shuffled. Each new implant in the study, at the time of surgery, after the cleaning and decontamination of the surface will be sorted for one treatment group. One envelope of subsequent numbering will be opened by a surgical assistant to determine the procedure that will be performed. In this way the individuals will be listed in each of the two different treatment groups.

Peri-implantitis treatment Individuals will be allocated at the time of surgery in each of the following treatment groups: Group 1: surgical debridement of the defect and mechanical decontamination by means of plastic curettes, bone defects will be treated later with JHS COL-HAP91® + JHS HAP-91® (n = 15); Group 2: only surgical debridement and mechanical decontamination by means of plastic curettes (n = 15). All groups will receive the same treatment for implant surface decontamination: debridement with plastic curette Implacare Hu-Friedy®, cleaning the surface with chlorhexidine gel 2% during 3 minutes and abundant irrigation with saline solution 0.9%.

All individuals should follow the following post operative drug protocol: use of Amoxicillin 500 mg 3 times a day for 07 days after surgery. Individuals allergic to Amoxicillin will be treated with Clindamycin 300 mg, 3 times a day, for 07 days. Analgesics, Tylenol 750 mg 3 times a day, and anti-inflammatory Nimesulide 100 mg 2 times a day will be prescribed.

Oral hygiene care will be strengthened and will be prescribed mouthwash two times a day (12/12 hour) 0.12% chlorhexidine during 21 days. Postoperative control will be carried out with 5, 10, 15 and 30 days. Return and maintenance shall be carried out with 60 and 90 days, at these moments new clinical examination will be held to evaluate peri-implant conditions, reinforcement for oral hygiene and prophylaxis. Recall visits with 6, 12 and 18 months will be made to measure peri-implant and maintenance parameters.

Standardized radiographic examinations will be carried out previously to the surgery, immediately after the surgery and with 6, 12 and 18 months for assessment of changes in bone levels obtained with the surgical procedures. Through comparison and measures carried out with x-rays performed preoperatively benchmarks as tops and valleys of the threads and the head of the implants will be used to carry out the measurements.

The x-rays will default on the exposure time and the positioning of the radiographic taking. Positioners and records will be used with dense silicone bite for standardization of survey position.

Peri-implant mucositis diagnosis An implant will be diagnosed with peri-implant mucositis in the presence peri-implant bleeding probing without bone loss.

Peri-implantitis diagnosis An implant will be diagnosed with peri-implantitis when present bleeding on probing and/or suppuration, a probing depth (PDi) greater than or equal to 5 mm and presence of bone loss confirmed by radiography, or a value of PDi greater than or equal to 5 mm even in the absence of bleeding or suppuration but presence of bone loss after radiographic examination.

The implants that shows PDi greater than or equal to 5 mm with bleeding on probing and not present bone loss, confirmed by radiographic examination, will be diagnosed as peri-implant mucositis and will not be included in the study.

Determination of peri-implant clinical status The following clinical parameters will be evaluated and recorded for all implants present in the oral cavity, with the exception of bone loss that will meet specific criteria (only implants with clinical signs of peri-implantitis): Plaque Index (PIi) (Silness and Löe, 1964 modified by Mombelli et al. 1987) (26, 27); Peri-implant probing depth in millimeters (PPDi); % os sites with peri-implant bleeding on probing (BOPi); Peri-implant suppuration (absence or presence) (Si); The presence and amount of peri-implant keratinized mucosa (KMi) (28); Presence of peri-implant bone loss in radiographic examination (BL).

Determination of radiographic bone level peri-implant Evaluation of peri-implant bone level will be held through periapical x-rays taken at the time of the examination of individuals by parallelism or standardized cone along with use of radiographic film positioners and acrylic bite records for standardization of position of the radiographic taking. Immediately after the surgical treatment, will be carried out x-rays and after 6, 12 and 18 months.

Evaluation of postoperative radiographic measurements must be carried out by another examiner, which does not have knowledge of the surgical treatment that was performed. Measures will be undertaken to assessment of post-treatment bone changes. For this it will be used as reference points the base of the platform and the turns of the implant.

Data of interest Through the assessment of individuals' records, shall be noted the following data concerning implants: implant installation time in months; amount of installed implants; implant function time in months; reason for tooth loss; periodontal phenotype (thin or thick); evaluation of occlusal functionality, type of the implants, implant surface treatment (present/absent) and when available type of surface treatment.

Clinical periodontal status The following clinical parameters will be evaluated and recorded for all teeth present in the oral cavity: Plaque Index (PIi) (Silness and Löe, 1964)(27); Pocket probing depth (PPD); Clinical attachment level (CAL); % of sites with periodontal bleeding on probing (BOP).

ELIGIBILITY:
Inclusion Criteria:

* It will include individuals diagnosed with early to moderate peri-implantitis (probing depth between 5 and 10 mm) rehabilitated with implant supporting fixed prosthesis for at least 6 months. Due to the great variation in implants' length the probing depth can shows great variability. In this way it is complicated to establish a cutoff point to define the severity of the disease. So in order to minimize this limitation, the peri-implant bone defect should be angular or circular involving at least 3 threads and should not exceed 50% of the total length of the implant.

Exclusion Criteria:

* Smokers
* Individuals with blood glucose more than 120 mg/dl or Insulin dependent diabetes
* Individuals who have undergone treatment of peri-implant disease over the last 6 months
* Individuals who used antibiotic therapy, for any reason, in the last 3 months
* Individuals who have any systemic condition that prevents surgical treatment
* Refusal to sign the informed consent
* A history of local radiotherapy to the head and neck region
* Pregnancy and lactation
* Active, uncontrolled periodontal pathology of the remaining dentition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Changes in peri-implant probing depth | one year and half. Pre-operative, after surgery: 6, 12 and 18 months
  Peri-implant probing depth measured in millimeters with peri-implant probe

SECONDARY OUTCOMES:
Changes in radiographic marginal bone level on standardized intraoral radiographs | One year and half. Pre operative and after surgery: immediatelly, 6, 12 and 18 months
  Evaluation of peri-implant bone level will be held through periapical x-rays taken at the time of the examination of individuals by parallelism or standardized cone along with use of radiographic film positioners and acrylic bite records for standardization of position of the radiographic taking.

OTHER OUTCOMES:
Presence of bleeding on probing | One year and half. Before treatment and after 6, 12, 18 months post surgery
  % os sites with peri-implant bleeding on probing

CONTACTS AND LOCATIONS:
Overall Officials: Sergio D Ferreira, MsC, Principal Investigator — Doctoral student
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil